CLINICAL TRIAL: NCT01144195
Title: An Open-label, Phase II Clinical Trial of Panitumumab in Combination With FOLFIRI Chemotherapy as Second Line Treatment in Subjects With Metastatic Colorectal Cancer Expressing Wild-type KRAS and Who Had Progressed ≥ 6 Months After the Last Dose of the First Line Chemotherapy
Brief Title: A Clinical Trial of Panitumumab in Combination With FOLFIRI Chemotherapy as Second Line Treatment in Subjects With Metastatic Colorectal Cancer Expressing Wild-type KRAS and Who Had Progressed ≥ 6 Months After the Last Dose of the First Line Chemotherapy
Acronym: ACTIVE
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Associacio catalana per a la recerca oncologica i les seves implicacions sanitaries i socials (Other)
Collaborators: Amgen (Industry)
Responsible Party: Dra. Inmaculada Portal, Associacio catalana per a la recerca oncologica i les seves implicacions sanitaries i socials
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACROSS-08-01; 2009-010975-26 (EudraCT Number)
Record Dates: First submitted 2010-06-07; First posted 2010-06-15 (Estimated); Last update posted 2010-11-10 (Estimated); Status verified 2010-11

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Panitumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Panitumumab + FOLFIRI — Panitumumab will be administered by intravenous (IV) infusion at a dose of 6 mg/kg once every 2 weeks. FOLFIRI chemotherapy will be administered once every 2 weeks after the administration of Panitumumab.

SUMMARY:
First line chemotherapy treatment regimens for metastatic colorectal cancer (mCRC) present disease-free survival of more than 10 months, and as much as 12 and 15 months for many patients.

It is evident that there are 2 groups of patients with metastatic colorectal cancer(mCRC): those who progress during first line treatment or in the 6 months following the last chemotherapy infusion and those who progress after this first 6-month period.

There are currently no studies evaluating the efficacy of second line chemotherapy regimens according to the duration of response to first line treatment. It seems logical that patients with less aggressive tumours will benefit more from treatments targeting specific proteins, such as panitumumab, due to the shorter duration of these tumours cell cycle, which makes them less sensitive to chemotherapy.

This study is therefore justified to determine an increase in activity and control of the disease in patients who progressed after 6 months of the last first line chemotherapy infusion for metastatic colorectal cancer(mCRC) in subjects expressing wild-type KRAS.

DETAILED DESCRIPTION:
This is a Phase II, single-arm, multi-centre study. Patients with metastatic colorectal cancer expressing wild type KRAS will be screened for this trial. KRAS mutation status will be assessed before inclusion and only WILD-TYPE-KRAS subjects will be included. Eligible subjects will be enrolled and treated with combination therapy consisting of Panitumumab and FOLFIRI as second line treatment.

Eligible patients must not have progressed on or within 6 months after receiving first line chemotherapy based on fluoropyrimidines and oxaliplatin (prior adjuvant chemotherapy based on fluoropyrimidine is permitted). Only one previous chemotherapy regimen is permitted. Progression after 6 months receiving first line chemotherapy regimen, should be imaging-based.

Tumor response assessment will be performed by the investigator per the modified Response Evaluation Criteria in Solid Tumors (m-RECIST). Subjects will be evaluated for tumor response every 6 weeks ± 1 week the first 24 weeks and every 8 weeks thereafter (per the modified-RECIST criteria) until progression disease (PD) or withdrawal from the trial. Responding disease will be confirmed no less than 28 days after the criteria for response are first met. Subjects with symptoms suggestive of progression disease(PD) should be evaluated for tumor progression at the time the symptoms occur.

All subjects who permanently discontinue the treatment for any reason, will undergo a safety follow-up assessment 30 days ± 7 days after the last treatment dose Subjects will be followed for disease status and subsequent cancer therapy. All subjects who discontinue all the treatment before disease progression (eg, due to unacceptable toxicities) are followed for progression free survival (PFS) (eg, radiographic tumor assessments) every 12 weeks ± 14 days until disease progression or the end of study (unless the reason for study discontinuation is fully withdrawn consent). After disease progression, all subjects are followed every 12 weeks ± 14 days from the safety follow-up visit until the end of study (approximately 52 weeks after the last subject is enrolled).

ELIGIBILITY:
Inclusion Criteria:

* Men or women 18 years of age or older
* Competent to comprehend, sign, and date an Independent Ethics Committee (IEC)/Institutional Review Board (IRB)-approved informed consent form
* Adenocarcinoma of the colon or rectum confirmed histologically or cytologically by the investigator in subjects presenting metastatic disease
* Subjects with wild-type KRAS tumor status confirmed by central laboratory assessment of paraffin-embedded tumor tissue from the primary tumor or metastasis.
* Radiologically documented progression of the disease according to modified RECIST criteria, 6 months or more after the last dose of chemotherapy for mCRC.
* Only one previous chemotherapy regimen for mCRC, consisting of first line chemotherapy based on fluoropyrimidines and oxaliplatin (prior adjuvant chemotherapy based on fluoropyrimidine is permitted).
* At least 1 uni-dimensionally measurable lesion of at least 20 mm per modified RECIST criteria. (All sites of disease must be evaluated ≤ 28 days prior to enrollment)
* If subject has prior history of cancer other than colorectal carcinoma, basal cell carcinoma, or cervical carcinoma in situ, then subject must not have had treatment or active disease within 5 years.
* Karnofsky performance status ≥ 70% at the time of enrolment in the study.
* Life expectancy ≥ 3 months
* Prior radiotherapy is acceptable (target lesions should not have been irradiated). At least 14 days must have passed since the administration of the radiotherapy and all signs of early toxicity must have remitted.
* Haematological function (within the 7 days prior to starting the study treatment)::

  * Absolute Neutrophil Count(ANC) ≥ 1.5 x 109 cells/L
  * Hemoglobin ≥ 9.0 g/dL
  * Platelet count ≥ 100 x 109/L
* Kidney function (within the 7 days prior to starting the study treatment):

  * Creatinine ≤ 1.5 mg/dL
* Liver function (within the 7 days prior to starting the study treatment):

  * Aspartate Aminotransferase(AST) ≤ 3 x Upper Limit of Normal(ULN) (if liver metastases, ≤ 5 x ULN)
  * Alanine aminotransferase(ALT) ≤ 3 x ULN (if liver metastases, ≤ 5 x ULN)
  * Bilirubin ≤ 2 x ULN
* Metabolic function (within the 7 days prior to starting the study treatment):

  * Magnesium ≥ lower limit of normal Lower Limit of normal(LLN),
  * Calcium ≥ lower limit of normal (LLN)

Exclusion Criteria:

* More than one previous chemotherapy regimen for mCRC consisting of first line chemotherapy based on fluoropyrimidines and/or oxaliplatin (patients receiving first-line chemotherapy based on irinotecan are not candidate for this study).
* Progression of the disease during the first line treatment or less than 6 months after completing the last cycle of first line chemotherapy for mCRC.
* Systemic chemotherapy, hormone treatment, immune therapy or experimental or approved antibodies/proteins (e.g. bevacizumab) ≤ 30 days prior to inclusion.
* Unresolved toxicity from a prior systemic treatment which, in the investigator's opinion, makes the subject unsuitable for inclusion.
* Metastasis in brain/central nervous system (exception: subjects who have been treated, have asymptomatic metastases in the central nervous system and have not been receiving steroids for at least the 30 days prior to inclusion in the study are eligible).
* Significant cardiovascular disease, including unstable angina pectoris or myocardial infarction within the 6 months prior to the start of the study treatment, or history of ventricular arrhythmia.
* Previous treatment with anti-EGFr antibodies (e.g. cetuximab) or treatment with small molecule Epidermal Growth Factor Receptor (EGFr) tyrosine kinase inhibitors (e.g. erlotinib).
* History of interstitial pneumonia or pulmonary fibrosis or signs of interstitial pneumonia or pulmonary fibrosis on the baseline chest X-ray.
* Treatment for systemic infection within the 14 days prior to starting the study treatment.
* Radiotherapy ≤ 14 days prior to inclusion. Patients must have recovered from all radiotherapy-related toxicity.
* Active inflammatory bowel or other intestinal disease causing chronic diarrhoea (defined as > 4 loose bowel movements per day).
* History of Gilbert's syndrome or dihydropyrimidine deficiency.
* History of any disease which could increase the risks associated to participation in the study or interfere in the interpretation of the study results.
* Known positive test for infection by human immune deficiency virus, hepatitis C, chronic active hepatitis B.
* Subject allergic to the ingredients of the study medication of protein A of Staphylococcus.
* Any comorbid disease which could increase the risk of toxicity.
* The subject presents a disorder of any kind which compromises his/her ability to provide informed consent in writing and/or follow the study procedures.
* Any investigational agent within the 30 days prior to inclusion.
* Major surgery within the 28 days prior to study enrollment.
* Pregnant or breastfeeding women.
* Women or men of childbearing age who do not agree to use appropriate double barrier contraceptive methods (e.g. diaphragm plus condom) or remain abstinent throughout the study and for 6 months after the last administration of the study drug for women and 1 month for men.
* Subjects who do not wish to meet the study requirements or are unable to do so.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2009-09; Primary Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | 3 years

SECONDARY OUTCOMES:
disease control rate | 3 years
duration of response | 3 years
time to response | 3 years
progression-free survival | 3 years
time to progression | 3 years
time to treatment failure | 3 years
duration of stable disease | 3 years
Incidence of adverse events | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Carles Pericay, MD PhD, Study Chair — Corporació Sanitaria Parc Taulí, Sabadell (Spain); Ferran Losa, Dr., Principal Investigator — Hospital General de l'Hospitalet; Pilar Vicente, Dra., Principal Investigator — Hospital General de Granollers; Hermini Manzano, Dr., Principal Investigator — Hospital Son Dureta; Juan Manuel Campos, Dr., Principal Investigator — Hospital Arnau de Vilanova (Valencia); Joan Manel Gasent, Dr., Principal Investigator — Hospital de Denia; Enrique Barrajón, Dr., Principal Investigator — Clínica de Benidorm; Inma Guasch, Dra., Principal Investigator — Hospital General de Manresa; Antonia Salud, Dra., Principal Investigator — Hospital Arnau de Vilanova (Lleida); Miquel Nogué, Dr., Principal Investigator — Hospital General de Vic; Inés Cabezas, Dra., Principal Investigator — Hospital Sant Joan de Reus; Jordi Alfaro, MD, Principal Investigator — Consorci Sanitari de Terrassa
Locations (1):
- Associació Catalana per la Recerca Oncològica i les Seves Implicacions Sanitaries i Socials, Barcelona, Barcelona, Spain